CLINICAL TRIAL: NCT05639998
Title: Phase 2 Randomized, Multi-centric of Heterologus Prime-Boost Combination of SARS-CoV-2 Vaccines to Evaluate the Immunogenicity and Safety of BBV152 (COVAXIN®) With BBV154 (Adenoviral Intranasal COVID-19 Vaccine) in Healthy Volunteers
Brief Title: BBV152/BBV154 Heterologus Prime-Boost Study
Acronym: BBV152BBV154
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BBIL-BBV152/154-2021
Record Dates: First submitted 2022-08-17; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Group 1 (COVAXIN® + COVAXIN®): In this group, 152 participants will be recruited who will receive COVAXIN® on day 0 and on day 28 via the intramuscular route.
  Group 2 (COVAXIN® + BBV154): In this group, 152 participants will be recruited who will receive COVAXIN® (Intramuscular) on day 0 and BBV154 (Intranasal) day 28.
  Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® viaintramuscular route.
  Group 3 (BBV154 + COVAXIN®): In this group, 152 participants will be recruited who will receive BBV154 (Intranasal) on day 0 and COVAXIN® (Intramuscular) on day 28.
  Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® via intramuscular route.
  Group 4 (BBV154 + BBV154): In this group, 152 participants will be recruited who will receive BBV154 on day 0 and on day 28 via the intranasal route
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1(COVAXIN® + COVAXIN®) (Experimental): Group 1 (COVAXIN® + COVAXIN®):
  In this group, 152 participants will be recruited who will receive COVAXIN® on day 0 and on day 28 via the intramuscular route
  Interventions: Biological: COVAXIN(BBV152)
- Group 2(COVAXIN® + BBV154) (Experimental): Group 2 (COVAXIN® + BBV154):
  In this group, 152 participants will be recruited who will receive COVAXIN® (Intramuscular) on day 0 and BBV154 (Intranasal) day 28.
  *Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® via intramuscular route
  Interventions: Biological: COVAXIN(BBV152); Biological: BBV154 Intranasal Vaccine
- Group 3(BBV154 + COVAXIN®) (Experimental): Group 3 (BBV154 + COVAXIN®):
  In this group, 152 participants will be recruited who will receive BBV154 (Intranasal) on day 0 and COVAXIN® (Intramuscular) on day 28.
  *Post 56 days of vaccination, participants with sero-conversion rate less than 3 folds will receive another dose of COVAXIN® via intramuscular route
  Interventions: Biological: COVAXIN(BBV152); Biological: BBV154 Intranasal Vaccine
- Group 4(BBV154 + BBV154) (Experimental): Group 4 (BBV154 + BBV154):
  In this group, 152 participants will be recruited who will receive BBV154 on day 0 and on day 28 via the intranasal route.
  Interventions: Biological: BBV154 Intranasal Vaccine

INTERVENTIONS:
Biological: COVAXIN(BBV152) — COVAXIN® on day 0 and on day 28 via the intramuscular route in GROUP 1. COVAXIN® (Intramuscular) on day 0 and BBV154 (Intranasal) day 28:GROUP 2
  Arms: Group 1(COVAXIN® + COVAXIN®); Group 2(COVAXIN® + BBV154); Group 3(BBV154 + COVAXIN®)
Biological: BBV154 Intranasal Vaccine — BBV154 (Intranasal) on day 0 and COVAXIN® (Intramuscular) on day 28: GROUP 3 BBV154 on day 0 and on day 28 via the intranasal route: GROUP 4
  Arms: Group 2(COVAXIN® + BBV154); Group 3(BBV154 + COVAXIN®); Group 4(BBV154 + BBV154)

SUMMARY:
All participants will be assessed for immunogenicity and safety endpoints and provide a blood sample before the administration of the first dose of IP. Blood samples will be collected on days 0, 9 (Groups 1, 3 and 4), 28,37 (Groups 2 and 4), 56, 90 and 180 to assess the neutralizing antibody titer against the SARSCoV-2 virus. A subset of 160 Participants (40 participants from each group) will be assessed for immunogenicity analysis, among these subset 10mL of blood and 5mL of saliva will be collected on days 0, 9 (Groups 1, 3 and 4), 28, 37 (Groups 2 and 4), 56, 90 and 180 to assess cell-mediated immunity and mucosal immunogenicity.

Group 1 (COVAXIN® + COVAXIN®): In this group, 152 participants will be recruited who will receive COVAXIN® on day 0 and on day 28 via the intramuscular route.

Group 2 (COVAXIN® + BBV154): In this group, 152 participants will be recruited who will receive COVAXIN® (Intramuscular) on day 0 and BBV154 (Intranasal) day 28.

*Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® viaintramuscular route.

Group 3 (BBV154 + COVAXIN®): In this group, 152 participants will be recruited who will receive BBV154 (Intranasal) on day 0 and COVAXIN® (Intramuscular) on day 28.

*Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® via intramuscular route.

Group 4 (BBV154 + BBV154): In this group, 152 participants will be recruited who will receive BBV154 on day 0 and on day 28 via the intranasal route.

DETAILED DESCRIPTION:
A Phase 2 randomized, multi-centric, Clinical Trial of Heterologus Prime-Boost Combination of SARS-CoV-2 Vaccines to evaluate the immunogenicity and safety of BBV152 (COVAXIN®) with BBV154 (Adenoviral Intranasal COVID-19 vaccine) in Healthy Volunteers.

This is a heterologus prime boost study, designed to evaluate the immunogenicity and safety of COVAXIN® with BBV154 and vice versa, amongthe four groups. A total of 608 subjects will be enrolled in the 1:1:1:1 ratio.

Group 1 (COVAXIN® + COVAXIN®): In this group, 152 participants will be recruited who will receive COVAXIN® on day 0 and on day 28 via the intramuscular route.

Group 2 (COVAXIN® + BBV154): In this group, 152 participants will be recruited who will receive COVAXIN® (Intramuscular) on day 0 and BBV154 (Intranasal) day 28.

*Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® viaintramuscular route

Group 3 (BBV154 + COVAXIN®): In this group, 152 participants will be recruited who will receive BBV154 (Intranasal) on day 0 and COVAXIN® (Intramuscular) on day 28.

*Post 56 days of vaccination, participants with seroconversion rate less than 3 folds will receive another dose of COVAXIN® via intramuscular route.

Group 4 (BBV154 + BBV154): In this group, 152 participants will be recruited who will receive BBV154 on day 0 and on day 28 via the intranasal route.

All participants will be assessed for immunogenicity and safety endpoints and provide a blood sample before the administration of the first dose of IP. Blood samples will be collected on days 0, 9 (Groups 1, 3 and 4), 28, 37 (Groups 2 and 4),56, 90 and 180 to assess the neutralizing antibody titer against the SARS-CoV-2 virus. A subset of 160 Participants (40 participants from each group) will be assessed for cell mediated and mucosal immunogenicity analysis, among these subset 10mL of blood and 5mL of saliva will be collected on days 0, 9 (Groups 1, 3 and 4), 28, 37 (Groups 2 and 4), 56, 90 and 180 to assess cell-mediated immunity and mucosal immunogenicity.

STUDY PROCEDURE

Visit 1(Day 0)

* If the participant is eligible (in good general health or stable pre-existing disease as per the discretion of the Principal investigator), a blood sample will be withdrawn before vaccination for all the participants.
* Safety Labs: An additional 15mL of blood will collected from half of the study population (76 from each group) to assess the safety at Day 0 and 56.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment. A study vaccine/comparator will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes of observation to record any immediate adverse event.
* Additional 10 mL blood will be collected from subset of 160 participants (Group1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of 160 participants (Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* Vaccine will be administered.
* Diary cards will be distributed to the participants.
* Telephonic follow-up (1-7-days post-vaccination) for adverse event recording.

Visit 2 (Day 9+2):

* Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Subset of Study participants (Group 1, 3 and 4) will return to the OPD for vitals and physical examination (general and systemic examination), and specific symptoms for COVID-19.
* Additional 10 mL blood will be collected from subset of (Groups 1, 3 and 4)participants(Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of (Groups 1, 3 and 4) participants(Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).

Visit 3 (Day 28 +2 ):

* Study participants will return to the OPD for vitals and physical examination (general and systemic examination), and specific symptoms for COVID-19.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Additional 10 mL blood will be collected from subset of 160 participants(Group1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected fromsubset of 160 participants(Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* Vaccine will be administered.
* Telephonic follow-up (1-7-days post-vaccination) for adverse event recording.

Visit 4 (Day 37±2):

* Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Subset of Study participants (Groups 2 and 4) will return to the OPD for vitals and physical examination (general and systemic examination), and specific symptoms for COVID-19.
* Additional 10 mL blood will be collected from subset of (Groups 2 and 4) participants (Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of (Groups 2 and 4) participants (Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).

Visit 5 (Day 56+7):

* Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
* Safety Labs: 15mL of blood will collected from half of the study population (76 from each group) to assess the safety.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Additional 10 mL blood will be collected from subset of 160 participants(Group1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of 160 participants (Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).

Visit 6 (Day 90+7):

* Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Additional 10 mL blood will be collected from subset of 160 participants(Group1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of 160 participants(Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).

Visit 7 (Day 180+7):

* Study participants will return to the OPD for physical examination (general and systemic examination), and specific symptoms for COVID-19.
* A blood sample (5 mL) will be collected from all the participants for immunogenicity assessment.
* Additional 10 mL blood will be collected from subset of 160 participants (Group1:40, Group-2:40, Group 3: 40 and Group 4: 40).
* A 5mL saliva sample will be collected from subset of 160 participants (Group-1:40, Group-2:40, Group 3: 40 and Group 4: 40).

DSMB & report

An interim report based on the safety and immunogenicity of the vaccineswill be notified to the Data safety monitoring board and Central Drugs Standard Control Organization (CDSCO), India, for further progressing theclinical development of the vaccine. This interim report will contain a detailed analysis of the data based on the primary and secondary objectives through Day 56 (Immunogenicity & Safety).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Participants of either gender, ages between 18 years <65 Years.
3. Good general health as determined by the discretion of investigator (vital signs (heart rate 60 to 100 bpm; blood pressure systolic 90 mm Hg and <140 mm Hg; diastolic 60 mm Hg and <90 mm Hg; oral temperature <100.4ºF), medical history, and physical examination).
4. Expressed interest and availability to fulfil the study requirements.
5. For a female participant of child-bearing potential, planning to avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least four weeks after the last vaccination
6. Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner from first vaccination until 3 months after last vaccination .
7. Participants must refrain from blood/plasma or any other bodily fluid donation from the time of first vaccination until 3 months after the last vaccination
8. Agrees not to participate in another clinical trial at any time during the study period.
9. Agrees to remain in the study area for the entire duration of the study.
10. Willing to allow storage and future use of biological samples for future research

Exclusion Criteria:

1. History of any other COVID-19 investigational/or licensed vaccination.
2. History of cold, sneezing, nasal obstruction in the past 1 day.
3. For women of childbearing potential, a positive urine pregnancy test (within 24 hours of administering each dose of vaccine).
4. Temperature >38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within three days before each dose of vaccine.
5. Medical problems because of alcohol or illicit drug use during the past 12 months.
6. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrolment or expects to receive an investigational agent during the study period.
7. Receipt of any licensed vaccine within four weeks before enrolment in this study.
8. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
9. Receipt of immunoglobulin or other blood products within the three months before vaccination in this study.
10. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
11. Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (nasal and topical steroids are allowed).
12. Any history of anaphylaxis concerning vaccination.
13. History of any cancer.
14. History of severe psychiatric severe conditions likely to affect participation in the study.
15. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venipuncture.
16. Any other serious chronic illness requiring immediate hospital specialist supervision.
17. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol. Re-Vaccination Exclusion Criteria
18. Pregnancy.
19. Anaphylactic reaction following administration of the vaccine.
20. Virologically confirmed cases of SARS-CoV-2 infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
immunogenicity | Day 0
  GMT and four-fold seroconversion rate (SCR) of neutralizing antibodies (NAb's) by MNT/PRNT assays across the four groups.
immunogenicity | Day 28+2
  GMT and four-fold seroconversion rate (SCR) of neutralizing antibodies (NAb's) by MNT/PRNT assays across the four groups
immunogenicity | Day56±7
  GMT and four-fold seroconversion rate (SCR) of neutralizing antibodies (NAb's) by MNT/PRNT assays across the four groups.
immunogenicity | Day90±7
  GMT and four-fold seroconversion rate (SCR) of neutralizing antibodies (NAb's) by MNT/PRNT assays across the four groups.
immunogenicity | Day180 ±7
  GMT and four-fold seroconversion rate (SCR) of neutralizing antibodies (NAb's) by MNT/PRNT assays across the four groups.

SECONDARY OUTCOMES:
reactogenicity | within 30 minutes post each vaccination
  The occurrence of immediate adverse events
immediate adverse events | within 30 minutes post each vaccination
  The occurrence of immediate adverse events
reactogenicity | within seven days of vaccination
  The occurrence of solicited adverse events
solicited adverse events | within seven days of vaccination
  The occurrence of solicited adverse events
reactogenicity | throughout the study duration 7 Months
  The occurrence of serious adverse events (SAEs)
serious adverse events | throughout the study duration 7 Months
  The occurrence of serious adverse events (SAEs)
reactogenicity | Day 0 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
reactogenicity | Day 9 +2
  The occurrence of any unsolicited adverse events
reactogenicity | Day 28 +2
  The occurrence of any unsolicited adverse events
reactogenicity | Day 37±2
  The occurrence of any unsolicited adverse events
reactogenicity | Day 56+7
  The occurrence of any unsolicited adverse events
unsolicited adverse events | Day 0 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
unsolicited adverse events | Day 9 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
unsolicited adverse events | Day 28 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
unsolicited adverse events | Day 37 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
unsolicited adverse events | Day 56 from the 1st dose vaccination
  The occurrence of any unsolicited adverse events
vaccine-induced Cell mediated immune response (Subset n=160) | day 9+2 (Group 1, 3 and 4)
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups
vaccine-induced Cell mediated immune response (Subset n=160) | days 28+2
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups
vaccine-induced Cell mediated immune response (Subset n=160) | 37±2 (Group 2 and 4)
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups
vaccine-induced Cell mediated immune response (Subset n=160) | 56±7
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups
vaccine-induced Cell mediated immune response (Subset n=160) | day 90±7
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups
vaccine-induced Cell mediated immune response (Subset n=160) | Day 180±7.
  Vaccine-induced cell-mediated immunogenicity and antigen-specific T-cell responses across the groups

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - The INCLEN Trust International/Guru Nanak Hospital, Gurgaon, Haryana
  - JSS Medical College & Hospital, Mysore, Karnataka
  - Gillurkur Multispeciality Hospital, Nagpur, Maharashtra
  - All India Institute of Medical Scienecs, New Delhi, National Capital Territory of Delhi
  - Institute of Medical Sciences and SUM Hospital,Odisha, Bhubaneswar, Odisha
  - Malla Reddy Narayana Multispeciality Hospital, Hyderabad, Telangana
  - Gleneagles Global Hospitals,Hyderabad, Hyderabad, Telangana
  - St Theresas Hospital, Hyderabad, Telangana
  - Prakhar Hospital Pvt Limited, Kanpur, Uttar Pradesh
  - The Medicity Hopsital, Rudrapur, Uttarakhand
  - Institute of Liver and Biliary Sciences,New Delhi, Delhi